CLINICAL TRIAL: NCT05641532
Title: Physical Activity Intervention for Persons Newly Diagnosed With Multiple Sclerosis
Brief Title: Physical Activity in Persons Newly Diagnosed With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elizabeth Barstow, Faculty Advisor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300009893
Record Dates: First submitted 2022-11-14; First posted 2022-12-07 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Physical activity; Newly diagnosed with MS; Behavior change; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will undergo one intervention condition remotely delivered using electronic newsletters and one-on-one video coaching. Outcome measures will be assessed at two time points: baseline and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capability-Opportunity-Motivation-Behavior (COM-B) based physical activity behavioral intervention (Experimental): This is a 1-arm study with an intervention condition based on the COM-B model
  Interventions: Behavioral: Physical activity behavioral intervention in persons newly diagnosed with MS

INTERVENTIONS:
Behavioral: Physical activity behavioral intervention in persons newly diagnosed with MS — 1. The newsletters will provide the knowledge, skills, resources, and strategies for promoting physical activity in persons newly diagnosed with MS. These newsletters will be released seven times during the program. The first three newsletters will be released weekly, and the last four will be released every other week.
  2. The one-on-one video coaching chats with participants will be conducted via Zoom, which consist of discussion and elaboration of newsletters content, supportive accountability, feedback and encouragement on behavior change. The chats further provide social persuasion for promoting behavior change. The chats are semi-scripted and individualized interventions (~15 - 30 minutes/chat). The chats will occur seven times during the week when a newsletter is delivered.
  3. The intervention includes a pedometer (NL-800 pedometer), a logbook, and a calendar for tracking daily step counts, planning of physical activity, setting goals, and monitoring progress over the program.

SUMMARY:
This single group pre-post pilot intervention will examine the feasibility and initial effect of a 12-week behavioral intervention, based on the Behavior Change Wheel and Capability-Opportunity-Motivation-Behavior (COM-B) model and remotely delivered through electronic newsletters and online one-on-one video conferencing, for promoting physical activity and secondarily reducing fatigue and quality of life in persons newly diagnosed with MS (diagnosed with MS within the past 2 years). The investigators hypothesize the proposed 12-week intervention will be feasible based on process, resource, management, and scientific outcomes. The investigators further hypothesize that individuals who receive the 12-week intervention will demonstrate an increase in physical activity behavior, particularly daily step counts, and reduce fatigue.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Diagnosed with multiple sclerosis for 2 or fewer years
* Fully ambulatory
* No relapse within the last 30 days
* Non-active (Godin Leisure-Time Exercise Questionnaire - Health Contribution Score < 14)
* Able to read 14-point font size
* Internet & video conferencing access
* Undergoing disease-modifying therapy

Exclusion Criteria:

* Pregnancy
* Moderate or high risk for undertaking physical activity (≥ 2 affirmatives on the Physical Activity Readiness Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Feasibility metric: Process | 12 weeks
  Process assesses participant recruitment, retention, and adherence i. Recruitment and refusal rates ii. Retention, attrition, and adherence rates to study procedures
Feasibility metric: Resource | 12 weeks
  We will assess the resources required for the study.
Feasibility metric: Management | 12 weeks
  Management assesses data management.
Feasibility metric: Overall safety | 12 weeks
  Overall safety will be assessed through the number of adverse events.
Change of Physical Activity levels through Accelerometry from baseline and 12 weeks | 12 weeks
  Physical activity will be assessed using an ActiGraph accelerometer. Participants will wear an accelerometer on a belt around their waist during the waking hours of a 7 day period. Participants will complete this at baseline and 12 weeks
Change of Physical Activity levels through the Godin Leisure-Time Exercise Questionnaire from baseline and 12 weeks | 12 weeks
  Physical activity will be assessed using the Godin Leisure-Time Exercise Questionnaire. Participants will complete this questionnaire at baseline and 12 weeks.
Change of Physical Activity levels through the Abbreviated International Physical Activity Questionnaire from baseline and 12 weeks | 12 weeks
  Physical activity will be assessed using the Abbreviated International Physical Activity Questionnaire. Participants will complete this questionnaire at baseline and 12 weeks.

SECONDARY OUTCOMES:
Change of self-report measures of Fatigue through the Fatigue Severity Scale from baseline and 12 weeks | 12 weeks
  Self report measures of fatigue will be assessed through the Fatigue Severity Scale. Participants will complete this questionnaire at baseline and 12 weeks
Changes of self-report measures of quality of life through the Multiple Sclerosis Impact Scale-29 at baseline and 12 weeks | 12 weeks
  Self report measures of quality of life will be assessed through the Multiple Sclerosis Impact Scale-29.Participants will complete this questionnaire at baseline and 12 weeks
Formative evaluation | 12 weeks
  Participants' satisfaction in the study will be assessed through a self-developed survey which will be completed at 12 week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No